CLINICAL TRIAL: NCT06881719
Title: Training of Executive Functions Through the APP "The Apollo & Rosetta Adventures"
Brief Title: Experimental Research on the Training of Executive Functions Through the APP "The Apollo & Rosetta Adventures" (E-FAR) in Children with ADHD (8-13 Yrs)
Acronym: E-FAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Collaborators: IRCCS Eugenio Medea (Other)
Responsible Party: Principal Investigator, Gian Marco Marzocchi, Associate Professor, University of Milano Bicocca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PsicoMilanoBicocca
Record Dates: First submitted 2025-02-03; First posted 2025-03-18 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: ADHD
Keywords: EXECUTIVE FUNCTION; TRAINING; APP MOBILE
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Comparison of the effects of the App Apollo & Rosetta on Executive Function (EF) in a group of children with ADHD, compared to the typical development of EF in a group of children with ADHD not treated.
Who Masked: Investigator
Masking Description: Collaborators of the investigator are blind about the two groups (trained vs not-trained) when administering the tasks before and after the training
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Training Executive Function through Apollo and Rosetta app (Experimental): The new APP "The Adventures of Apollo and Rosetta" consists of 7 exercises The training program provides for the application of 36 mini-game sessions lasting 15-20 minutes each (alternating the first 4 and the last 3 games) over 12 weeks (the child must practice 3 times a week).
  Interventions: Device: The Adventures of Apollo & Rosetta
- Control group (No Intervention): A control group of children with ADHD with similar characteristics in terms of gender, age, IQ and severity of symptoms will be identified. The children in the control group will not undergo any therapy and will be tested before and after a 3-month interval.

INTERVENTIONS:
Device: The Adventures of Apollo & Rosetta — The new APP "The Adventures of Apollo and Rosetta" consists of 7 exercises (1. Explorer; 2. Deciphering codes; 3. Particle accelerator tunnel; and 4. Leaping asteroids, - 5. Galactic art; 6. Stellar Laboratory; 7. Challenge of opposites).
  The training program provides for the application of 36 mini-game sessions lasting 15-20 minutes each (alternating the first 4 and the last 3 games) over 12 weeks (the child must practice 3 times a week).
  The training via APP can be administered in the first sessions on an outpatient basis, then it can be delegated to parents who take care of the exercises 3 times a week (20-15-20 minutes). A work diary will be kept monitoring the progress of the activities.
  Arms: Training Executive Function through Apollo and Rosetta app

SUMMARY:
ADHD is one of the most prevalent neurodevelopmental disorders, with a strong impact on general functioning and in daily life. Executive Functions play an important role on this disorder, and numerous treatments have been developed over the years to try to contain its symptoms. The present study aimed to investigate whether the use of a video game, "The incredible adventures of Apollo and Rosetta", could enhance Fxecutive Functions and improve the impact of symptoms in children with ADHD. A longitudinal study was carried out with 35 subjects aged 8 to 11 years. They were assessed twice, at the beginning and after three months. 17 subjects were assigned to the experimental group, which downloaded and used the application systematically. 18 participants, on the other hand, were assigned to the wait-and-see condition, as a control group. Participants were administered four tests, while in contemporary, parents filled out two self-report questionnaires. A mixed between and within ANOVA was used to analyze the data. The results, although not showing significantly impactful effects, are promising and move in the direction of the research hypothesis. In fact, systematic use of this application appears to play a role in increasing executive functions and seems to act as a protective factor against any worsening.

DETAILED DESCRIPTION:
Introduction Executive Functions represent a series of coordinated and higher-order processes to allow the child to develop adequate self-regulation of behavior in order to implement adaptive behaviors. Executive deficits represent the most critical area in the 5-10 age group precisely because the development deficit of the prefrontal regions prevents the acquisition of skills which are then fundamental throughout the development to young adulthood.

The enhancement of Executive Functions for many children with atypical development is necessary to reduce subsequent developmental risks. Among the various training proposals, those that involve cognitive and motor processes are those that have shown the greatest benefits; it is also important that the child is motivated and experiences pleasure in carrying out these activities.

The use of APPs on tablets and computer games allows children to increase their motivation to play, eliciting the pleasure of doing fun exercises. The motivation to carry out the task allows the child to spend more time carrying out training to enhance Executive Functions and determines an improvement in cognitive skills.

The research group of the University of Feevale (Brazil) coordinated by Prof. Debora Nice Ferrari Barbosa has also created a new APP that stimulates Executive Functions in children, as demonstrated by their recent study on typical development. The video game is called "The adventures of Apollo and Rosetta" in which two characters face various missions in space in which they must avoid dangers or hit threatening objects according to the rules that are made explicit. The child must learn to remember rules, targets (working memory), stop automatic responses and manage distractions (inhibition) or change behavior patterns (flexibility).

The aim of the study is to verify whether the application of training via APP allows children with ADHD to improve performance in their Executive Functions and whether these improvements are generalized by reducing the symptoms of inattention and impulsivity.

Participants Participants in the study are 15 children with ADHD (in the absence of comorbidities) according to the ICD-10 criteria aged between 6 and 10 years who are not receiving any therapy (psychological and pharmacological) for the entire duration of the training (3 months). Diagnostic confirmation will occur through the administration of Conners-3 questionnaires (cut-off T> 65 of inattention and / or hyperactivity-impulsivity symptoms).

In addition to the experimental group, a control group of children with ADHD with similar characteristics in terms of gender, age, IQ and severity of symptoms will be identified. The children in the control group will not undergo any therapy and will be tested before and after a 3-month interval. Participants with ADHD from the experimental and control groups will be recruited at the IRCCS E. Medea in Bosisio Parini (LC).

Training The new APP "The adventures of Apollo and Rosetta" consists of 7 exercises (1. Explorer; 2. Deciphering codes; 3. Particle accelerator tunnel; and 4. Leaping asteroids, - 5. Galactic art; 6. Stellar Laboratory; 7. Challenge of opposites).

The training program provides for the application of 36 mini-game sessions lasting 15-20 minutes each (alternating the first 4 and the last 3 games) over 12 weeks (the child must practice 3 times a week).

The training via APP can be administered in the first sessions on an outpatient basis, then it can be delegated to parents who take care of the exercises 3 times a week (20-15-20 minutes). A work diary will be kept monitoring the progress of the activities.

Measures To verify the effectiveness of the intervention, behavioral measures are collected, before and after the training.

Primary outcome - Neuropsychological Tests:

1. Raven colored matrices to monitor Fluid Reasoning
2. the Ranette test of the BIA-R (Marzocchi et al, 2021) to evaluate the response inhibition capacity (administration in paper format);
3. the Horn Test (Marzocchi et al, 2013) to evaluate response inhibition and flexibility (using the "Self-regulate attention" software installed on a PC provided by the Milano-Bicocca University);
4. the Nepsy-II inhibition test (Korkman et al, 2007) to evaluate flexibility (administration in paper format);
5. the CO-TT test by Marsura et al (2020) to evaluate the updating component of working memory (the presentation of the items of this test will take place via power point, while the answers will be recorded on a paper protocol).

Secondary measures - Questionnaires:

1. Questionnaire for the assessment of executive functions (QUFE) - teachers and parents' version
2. Conners-3 Questionnaire to Assess ADHD Symptoms - Teachers and Parents Version.

Expected results It is hypothesized that ADHD children of the experimental group will improve their skills related to Executive Functions (near transfer) by finding a greater number of correct answers to the computerized tests. The improvement can be estimated in the measure of an effect size between 0.4 and 0.8 (average effect). Furthermore, a generalization of the improvements detected by the QUFE and Conners-3 questionnaires of about 0.3-0.4 (medium-low, but significant effect) is expected.

ELIGIBILITY:
Inclusion Criteria: Diagnosis of ADHD

Exclusion Criteria: Other neurodevelopmental disorder

-

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Executive Function and Attention tasks | 12 months
  To verify the effectiveness of the intervention, neuropsychological measures are collected, before and after the training.
  1. the number of correct responses at Ranette test of the BIA-R (Marzocchi et al, 2021) to evaluate the response inhibition capacity (administration in paper format);
  2. the decreased number of commission errors and the Reaction Time of correct responses at Horn Test (Marzocchi et al, 2013) to evaluate response inhibition and flexibility ;
  3. the number of correct responses at Nepsy-II inhibition test (Korkman et al, 2007) to evaluate flexibility (administration in paper format);
  4. the number of correct responses at CO-TT test by Marsura et al (2020) to evaluate the updating component of Working Memory.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS E. Medea, Bosisio Parini, Lecco
  - University of Milan Bicocca, Milan, Michigan

IPD SHARING:
Plan to Share IPD: Undecided